CLINICAL TRIAL: NCT00050583
Title: Treatment of Somatization in Primary Care
Brief Title: Treatment of Medically Unexplained Physical Ailments (Somatization Disorder)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Javier I Escobar MD, Associate Dean for Global Health, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH060265 (NIH); R01MH060265 (NIH)
Record Dates: First submitted 2002-12-16; First posted 2002-12-17 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Somatoform Disorders
MeSH Terms: conditions — Somatoform Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 10 Session modified CBT (including a relaxation component) administered by trained mental health clinicians at the primary care setting
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: CBT
- 2 (No Intervention): "Treatment as Usual", defined as the use of a consultation letter and traditional primary care management.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Ten Weekly Sessions of Manualized CBT
  Arms: 1
Behavioral: CBT — Cognitive Behavioral Therapy
  Arms: 1

SUMMARY:
The purpose of this study is to compare cognitive behavior therapy (CBT) to medical care-as-usual for the treatment of patients with high levels of medically unexplained physical symptoms (Somatization Disorder). A second goal is to examine the effectiveness of CBT in Latinos, since Latinos suffer a relatively high prevalence of Somatization Disorder.

DETAILED DESCRIPTION:
Patients with Somatization Disorder suffer from medically unexplained physical ailments and experience significant distress and disability. This disorder is an important problem for the primary health care system because patients with Somatization Disorder use health care resources extensively but receive little benefit. To date, no medical or psychiatric intervention has been demonstrated in controlled trials to produce clinically significant and lasting symptom relief or improved functional status in Somatization Disorder patients.

Patients in primary care settings with multiple unexplained symptoms are treated with 10 weekly sessions of CBT or "treatment as usual." Physical symptoms, comorbid psychiatric symptoms, disability, and health care utilization are measured and assessed through a combination of structured interviews and self-reports. Assessments are performed at study start, mid-treatment, end of treatment, and at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Somatization disorder

Exclusion Criteria:

* Bipolar disorder
* Schizophrenia or other psychosis
* Major Depression

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2001-02; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
CGI Improvement | Post Treatment

SECONDARY OUTCOMES:
Hamilton Depression | Post Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Javier I Escobar, M.D., Principal Investigator — Rutgers, The State University of New Jersey; Michael A Gara, Ph.D., Study Director — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ- Robert Wood Johnson Medical School; Dept. of Psychiatry, Piscataway, New Jersey, United States

REFERENCES:
- [Background] Escobar JI, Gara MA, Diaz-Martinez AM, Interian A, Warman M, Allen LA, Woolfolk RL, Jahn E, Rodgers D. Effectiveness of a time-limited cognitive behavior therapy type intervention among primary care patients with medically unexplained symptoms. Ann Fam Med. 2007 Jul-Aug;5(4):328-35. doi: 10.1370/afm.702. PMID 17664499